CLINICAL TRIAL: NCT02214420
Title: Simeprevir (SMV) + Sofosbuvir (SOF) With or Without Ribavirin (RBV) for Interferon-intolerant or Ineligible (IFN-II) Patients With Chronic Hepatitis C (CHC)
Brief Title: SMV + SOF With/Without RBV for IFN-II Patients With CHC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: SC Liver Research Consortium, LLC (Other)
Collaborators: Janssen, LP (Industry)
Responsible Party: Principal Investigator, Paul J. Pockros, MD, Principal Investigator, SC Liver Research Consortium, LLC
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PJPIIS-01-14
Record Dates: First submitted 2014-08-08; First posted 2014-08-12 (Estimated); Results first posted 2018-05-17 (Actual); Last update posted 2018-06-19 (Actual); Status verified 2018-05

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — Simeprevir; Sofosbuvir; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SMV+SOF (Active Comparator): IFN-II patients will receive 12 weeks of OLYSIO (Simeprevir) (150mg QD) + SOVALDI (Sofosbuvir) (400mg QD)
  Interventions: Drug: Simeprevir; Drug: Sofosbuvir
- SMV+SOF+RBV (Active Comparator): IFN-II patients will receive 12 weeks of OLYSIO (Simeprevir) (150mg QD) + SOVALDI (Sofosbuvir) (400mg QD) + weight-based Ribavirin 1000-1200 mg/day
  Interventions: Drug: Simeprevir; Drug: Sofosbuvir; Drug: Ribavirin

INTERVENTIONS:
Drug: Simeprevir
Drug: Sofosbuvir
Drug: Ribavirin
  Arms: SMV+SOF+RBV

SUMMARY:
Prior trials have shown that many G1 CHC patients are ineligible or intolerant to pegylated (PEG)-based regimens due to prior severe side effects, worsening of cytopenias, exacerbation of underlying psychiatric disorders, or autoimmune disorders. These patients will not be candidates for treatment with the approvals of SMV and SOF in early 2014 due to the combination with PEG-regimens. Results of the COSMOS study suggest that these patients are likely to have excellent responses to SMV+SOF with or without RBV with 12 weeks of therapy, and that 24 weeks are unnecessary. This trial is designed to rapidly enroll and be completed in order to confirm this hypothesis.

ELIGIBILITY:
Inclusion Criteria:

1. Targeted at least 20% enrollment of patients with cirrhosis
2. Adults >/= age 18 years.
3. Active infection with hepatitis C virus (HCV) genotype 1
4. Must have health insurance that covers therapy with SOF+RBV
5. Female patients of childbearing age must have a negative pregnancy test prior to initiating therapy, use at least two effective methods of contraception during treatment, and undergo monthly pregnancy tests.
6. Patients must be either IFN-ineligible due to psychiatric, autoimmune, neurological, or other causes that are confirmed appropriate by the PI; OR,
7. IFN-intolerant due to flu-like symptoms, psychiatric problems, cytopenia or other causes deemed appropriate by the PI.

Exclusion Criteria:

1. Presence of HIV co-infection
2. Presence of hepatocellular carcinoma (HCC)
3. Prior organ transplantation
4. Any history of hepatic decompensation
5. Patients taking any of the following medications:

   * Anticonvulsants- Carbamazepine, Oxcarbazepine, Phenobarbital, or Phenytoin.
   * Anti-infectives-erythromycin, clarithromycin, or telithromycin.
   * Antifungals- systemic itraconazole, ketoconazole, posaconazole, fluconazole, or voriconazole.
   * Antimycobacterials- rifampin, rifabutin or rifapentine.
   * Corticosteroids- systemic dexamethasone.
   * Propulsives- Cisapride.
   * Herbals- Milk thistle or St. John's Wart.
6. Patients that have been exposed to direct acting anti-viral agents
7. Patients with severe renal impairment (estimated Glomerular Filtration Rate (eGFR) <50 mL/min/1.73m2) or with end stage renal disease (ESRD).
8. Patients with platelet count <50 x109/L, Hemoglobin <10 g/dL, or Neutrophils <0.5 x109/L.
9. Women who are pregnant.
10. Men whose partners are pregnant or plan on becoming pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-10; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Pockros, MD, Principal Investigator — Scripps Clinic
Locations (3):
- United States (3):
  - Scripps Clinic, La Jolla, California
  - Icahn School of Medicine at Mt. Sinai, New York, New York
  - Clinical Research Centers of America, LLC, Murray, Utah

RESULTS

PARTICIPANT FLOW:
Groups:
- SMV+SOF: Interferon (IFN)-II patients will receive 12 weeks of OLYSIO (Simeprevir) (150mg QD) + SOVALDI (Sofosbuvir) (400mg QD)
  Simeprevir
  Sofosbuvir
- SMV+SOF+RBV: Interferon (IFN)-II patients will receive 12 weeks of OLYSIO (Simeprevir) (150mg QD) + SOVALDI (Sofosbuvir) (400mg QD) + weight-based Ribavirin 1000-1200 mg/day
  Simeprevir
  Sofosbuvir
  Ribavirin
Period: Overall Study
Arm/Group | SMV+SOF | SMV+SOF+RBV
Started | 14 | 10
Completed | 13 | 10
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- SMV+SOF: IFN-II patients will receive 12 weeks of OLYSIO (Simeprevir) (150mg QD) + SOVALDI (Sofosbuvir) (400mg QD)
  Simeprevir
  Sofosbuvir
- SMV+SOF+RBV: IFN-II patients will receive 12 weeks of OLYSIO (Simeprevir) (150mg QD) + SOVALDI (Sofosbuvir) (400mg QD) + weight-based Ribavirin 1000-1200 mg/day
  Simeprevir
  Sofosbuvir
  Ribavirin
- Total: Total of all reporting groups
Arm/Group | SMV+SOF | SMV+SOF+RBV | Total
Number analyzed (Participants) | 14 | 10 | 24
Age, Continuous [Mean (Full Range); unit: years] | 50.84 [22 to 76] | 58.31 [35 to 67] | 53.95 [22 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 3 | 12
  Male | 5 | 7 | 12
BMI [Mean (Full Range); unit: kg/m^2] | 29.47 [18.8 to 46.1] | 27.56 [19.1 to 42.9] | 28.67 [18.8 to 46.1]

OUTCOME MEASURES:

1. Primary Outcome: Sustained Viral Response
Description: Comparison of sustained virologic response at 12 weeks post-treatment (SVR12) in 2 arms of IFN-II patients: one receiving 12 weeks of simeprevir (SMV) (150mg QD)+ sofosbuvir (SOF) (400mg QD) and the second receiving to SMV (150mg QD)+SOF (400mg QD)+weight-based ribavirin (RBV) 1000-1200 mg/day. SVR12 is defined as a patient having undetectable hepatitis C virus (HCV) ribonucleic acid (RNA) levels 12 weeks post-treatment. Achieving SVR12 is generally indicative of hepatitis C infection being cured.
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | SMV+SOF | SMV+SOF+RBV
Number analyzed (Participants) | 14 | 10
Participants | 13 | 8

ADVERSE EVENTS:
Arm/Group | SMV+SOF | SMV+SOF+RBV
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/10
Other Adverse Events (participants affected / at risk) | 13/14 | 9/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SMV+SOF (N=14) | SMV+SOF+RBV (N=10)
Nausea or other GI discomfort (Gastrointestinal disorders) | 10 | 3
Fatigue (Nervous system disorders) | 5 | 4
Headache (Nervous system disorders) | 3 | 0
Cough and cold symptoms (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Photosensitivity (Skin and subcutaneous tissue disorders) | 2 | 0
Dizziness (Ear and labyrinth disorders) | 1 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Pruritis or rash (Skin and subcutaneous tissue disorders) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes